CLINICAL TRIAL: NCT06608134
Title: Safety and Feasibility of Umbilical Cord Wharton's Jelly Allograft Injections for
Brief Title: Safety and Feasibility of Umbilical Cord Wharton's Jelly Allograft Injections for Knee Osteoarthritis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: R3 Medical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R3-WJI-001
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis, Knee
Keywords: umbilical cord; Whartons Jelly; Allograft; knee pain; knee arthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: randomized, prospective, open label, dose escalation, non-controlled
Who Masked: Participant, Care Provider
Masking Description: With double blinding of the allograft neither participant nor provider will know what is being administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 2cc WJ Allograft (Low Dose) (Active Comparator): The 2cc Whartons Jelly Allograft group receives an intra-articular knee injection and is considered the Low Dose Group.
  Interventions: Biological: Umbilical Cord Wharton's Jelly Allograft Intra-articular Knee Injection
- 3cc WJ Allograft (Medium Dose) (Active Comparator): The 3cc Whartons Jelly Allograft group receives an intra-articular knee injection and is considered the Medium Dose Group.
  Interventions: Biological: Umbilical Cord Wharton's Jelly Allograft Intra-articular Knee Injection
- 4cc WJ Allograft (High Dose) (Active Comparator): The 4cc Whartons Jelly Allograft group receives an intra-articular knee injection and is considered the High Dose Group.
  Interventions: Biological: Umbilical Cord Wharton's Jelly Allograft Intra-articular Knee Injection

INTERVENTIONS:
Biological: Umbilical Cord Wharton's Jelly Allograft Intra-articular Knee Injection — Direct injection of biologic into the knee joint.

SUMMARY:
This is a Pilot Study which is randomized, prospective, open label, dose escalation, non-controlled evaluating safety and feasibility of intra-articular Wharton's Jelly (WJ) allograft will be evaluated in patients suffering with knee osteoarthritis. The participants will be randomized to one of three dosing treatment arms that will consist of one intra-articular knee injection containing either low dose, medium dose or high dose WJ allograft tissue.

DETAILED DESCRIPTION:
This is a Pilot Study which is randomized, prospective, open label, dose escalation, non-controlled study in which the safety and feasibility of intra-articular Wharton's Jelly (WJ) allograft will be evaluated in patients suffering with knee OA. The participants will be randomized to one of three dosing treatment arms that will consist of one intra-articular knee injection containing either low dose, medium dose or high dose WJ allograft tissue.

As this is a Pilot Study primarily designed to evaluate safety, no control will be used. The dosing groups will consist of either 2cc WJ Allograft (Low Dose), 3cc WJ Allograft (Medium Dose), or 4cc WJ Allograft (High Dose) with 120 total patients randomized into the three arms equally. In addition to baseline outcome instruments along with imaging and laboratory studies, patients will be followed for one year for evaluation of safety, pain relief and functional improvements.

ELIGIBILITY:
Inclusion Criteria:

* Be over age 30
* Diagnosed with Grade II or III OA on the KL scale (in one knee).
* Body Mass Index (BMI) <50Kg/m2
* Pain score of 4 or more on the Numeric Pain Rating Scale (NPRS)
* Female patients must be abstinent, surgically sterilized or postmenopausal
* Premenopausal females must have a negative pregnancy test, on contraceptive measures and do not anticipate pregnancy during the duration of the study.
* Be willing and capable of giving written informed consent to participate in English.
* Be willing and capable of complying with study-related requirements, procedures and visits in English.

Exclusion Criteria:

* Have taken any pain medication including nonsteroidal anti-inflammatory drugs (NSAIDs) within 2 weeks prior to study injection date.
* Use anticoagulants have a substance abuse history and fail to agree not to take any knee-symptom modifying drugs during the course of the study without discussing and reporting the use to the site principal investigator and study team.
* Have had an intra-articular injection of any drug including viscosupplementation in the index knee in the past 6 months.
* Have had surgery on the index knee with the past 6 months.
* Had a traumatic injury to the index knee with the past 3 months.
* Planned elective surgery during the course of the study.
* A history of organ or hematologic transplantation, rheumatoid arthritis, or other autoimmune disorders.
* Be on immunosuppressive medications.
* Have a diagnosis of carcinoma with the past 2 years.
* Have a knee infection or have used antibiotics for knee infection within the past 3 months.
* Have participated in any other clinical trial or treatment (not just for the knee, but for any reason) with any investigational product within the past 30 days prior to inclusion of study.
* Female patients who are breast feeding or are pregnant or desire to become pregnant during the course of the study.
* Contraindications to radiographic or MRI imaging.
* Serious neurological, psychological or psychiatric disorders.
* Injury or disability claims under current litigation or pending or approved workers compensation claims.
* Have a known drug allergy to amphotericin-B, ciprofloxacin, gentamycin, penicillin, or streptomycin.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
C Reactive Protein | Baseline, 1 week after the procedure, 6 weeks, 3 months, 6 months and one year
  C-reactive protein (CRP) is a protein made by the liver. The level of CRP increases when there's inflammation in the body. A simple blood test can check your C-reactive protein level.
  C-reactive protein is measured in milligrams per liter (mg/L). Results equal to or greater than 8 mg/L or 10 mg/L are considered high. Range values vary depending on the lab doing the test.
  A high test result is a sign of inflammation. It may be due to serious infection, injury or chronic disease. Your health care provider may recommend other tests to determine the cause.
Erythrocyte Sedimentation Rate | Baseline, 1 week after the procedure, 6 weeks, 3 months, 6 months and one year
  Sed rate, or erythrocyte sedimentation rate (ESR), is a blood test that can show inflammatory activity in the body.
  Because a sed rate test can't pinpoint the problem that's causing inflammation in your body, it's often accompanied by other blood tests, such as the C-reactive protein (CRP) test.
  ESR is measured in millimeters per hour (mm/hr). The normal values are:
  0 to 15 mm/hr in men 0 to 20 mm/hr in women
Alanine Transaminase | Baseline, 1 week after the procedure, 6 weeks, 3 months, 6 months and one year
  ALT is an enzyme that converts proteins into energy for the liver cells. Aspartate transaminase (AST). AST is an enzyme that helps the body break down amino acids. Alkaline phosphatase (ALP). ALP is an enzyme important for breaking down proteins. Albumin and total protein. Albumin is a protein made in the liver. Bilirubin. Bilirubin is a substance produced during the breakdown of red blood cells. Gamma-glutamyltransferase (GGT). Higher-than-usual may mean liver damage. L-lactate dehydrogenase (LD). LD is an enzyme found in the liver. Prothrombin time (PT). PT is the time it takes your blood to clot. Standard range:
  Alanine transaminase (ALT). ALT is an enzyme that converts proteins into energy for the liver cells. Standard range:
  ALT. 7 to 55 units per liter U/L.
Aspartate Transaminase | Baseline, 1 week after the procedure, 6 weeks, 3 months, 6 months and one year
  AST is an enzyme that helps the body break down amino acids. . Standard range: AST 8 to 48 units per liter
Alkaline Phosphatase | Baseline, 1 week after the procedure, 6 weeks, 3 months, 6 months and one year
  ALP is an enzyme important for breaking down proteins. Standard range: 40 to 129 units per liter
Albumin | Baseline, 1 week after the procedure, 6 weeks, 3 months, 6 months and one year
  Albumin is a protein made in the liver. Normal range is 34 to 54 grams/liter.
Creatinine | Baseline, 1 week after the procedure, 6 weeks, 3 months, 6 months and one year
  Creatinine is a waste product that comes from the digestion of protein in your food and the normal breakdown of muscle tissue. It is removed from the blood through your kidneys. Everyone has some creatinine in their blood, but too much can be a sign of a possible kidney problem. Normal range is 0.6-1.3 milligrams/deciliter
Blood Urea Nitrogen | Baseline, 1 week after the procedure, 6 weeks, 3 months, 6 months and one year
  blood urea nitrogen (BUN) test reveals important information about how well your kidneys are working. A BUN test measures the amount of urea nitrogen that's in your blood. Normal BUN is 6-20 milligrams/deciliter.

SECONDARY OUTCOMES:
36-Item Short Form Survey (SF-36) | Baseline, 24 hours after intervention, 1 week, 6 weeks, 3 months, 6 months, 1 year
  The SF-36 is used as an assessment tool to measure a quality of life. The SF-36 is comprehensive health survey with a total of 36 questions divided into eight categories, including physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). The score averages for each category range from 0 to 100, with a higher score defining a more favorable outcome.
Numerical Pain Rating Scale (NPRS) | Baseline, 24 hours after intervention, 1 week, 6 weeks, 3 months, 6 months, 1 year
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Knee Injury and Osteoarthritis Outcome Score | Baseline, 24 hours after intervention, 1 week, 6 weeks, 3 months, 6 months, 1 year
  This survey asks for your view about your knee. This information will help us keep track of how you feel about your knee and how well you are able to perform your usual activities.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - R3 Anti Aging Scottsdale, Scottsdale, Arizona
  - R3 Anti Aging Beverly Hills, Beverly Hills, California
  - Optimal Medical Group, Fresno, California
  - Scheer Medical Wellness, New York, New York
  - Dr. Duc (Steve) Le, MD, Cleveland, Texas

IPD SHARING:
Plan to Share IPD: Yes
R3 Medical Research will share study materials in a blinded fashion with no participant identifying information to participating researchers as needed.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Short term (6 months) and Long Term (12 months) for one month only.
Access Criteria: Secure, encrypted server.

REFERENCES:
- [Result] Cisternas MG, Murphy L, Sacks JJ, Solomon DH, Pasta DJ, Helmick CG. Alternative Methods for Defining Osteoarthritis and the Impact on Estimating Prevalence in a US Population-Based Survey. Arthritis Care Res (Hoboken). 2016 May;68(5):574-80. doi: 10.1002/acr.22721. PMID 26315529
- [Result] Van Manen MD, Nace J, Mont MA. Management of primary knee osteoarthritis and indications for total knee arthroplasty for general practitioners. J Am Osteopath Assoc. 2012 Nov;112(11):709-15. PMID 23139341
- [Result] Losina E, Thornhill TS, Rome BN, Wright J, Katz JN. The dramatic increase in total knee replacement utilization rates in the United States cannot be fully explained by growth in population size and the obesity epidemic. J Bone Joint Surg Am. 2012 Feb 1;94(3):201-7. doi: 10.2106/JBJS.J.01958. PMID 22298051
- [Result] Gupta A, Potty ASR, Ganta D, Mistovich RJ, Penna S, Cady C, Potty AG. Streamlining the KOOS Activities of Daily Living Subscale Using Machine Learning. Orthop J Sports Med. 2020 Mar 24;8(3):2325967120910447. doi: 10.1177/2325967120910447. eCollection 2020 Mar. PMID 32270015
- [Result] Farr J, Gomoll AH, Yanke AB, Strauss EJ, Mowry KC; ASA Study Group. A Randomized Controlled Single-Blind Study Demonstrating Superiority of Amniotic Suspension Allograft Injection Over Hyaluronic Acid and Saline Control for Modification of Knee Osteoarthritis Symptoms. J Knee Surg. 2019 Nov;32(11):1143-1154. doi: 10.1055/s-0039-1696672. Epub 2019 Sep 18. Erratum In: J Knee Surg. 2019 Nov;32(11):e2. doi: 10.1055/s-0039-3402742. PMID 31533151
- [Result] Hoorntje A, Witjes S, Koenraadt KLM, Aarts R, Weert T, van Geenen RCI. More Severe Preoperative Kellgren-Lawrence Grades of Knee Osteoarthritis were Partially Associated with Better Postoperative Patient-Reported Outcomes in TKA Patients. J Knee Surg. 2019 Mar;32(3):211-217. doi: 10.1055/s-0038-1635114. Epub 2018 Feb 28. PMID 29490401
- [Result] Kahn TL, Soheili A, Schwarzkopf R. Outcomes of total knee arthroplasty in relation to preoperative patient-reported and radiographic measures: data from the osteoarthritis initiative. Geriatr Orthop Surg Rehabil. 2013 Dec;4(4):117-26. doi: 10.1177/2151458514520634. PMID 24600532
- [Result] Eyichukwu GO. Non-Steroidal anti inflammatory drugs usage in orthopaedics and trauma practice. A guide and review. Niger J Med. 2010 Oct-Dec;19(4):374-81. doi: 10.4314/njm.v19i4.61959. PMID 21526623
- [Result] Yasir M, Goyal A, Sonthalia S. Corticosteroid Adverse Effects. 2023 Jul 3. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK531462/ PMID 30285357
- [Result] Gupta A, Woods MD, Illingworth KD, Niemeier R, Schafer I, Cady C, Filip P, El-Amin SF 3rd. Single walled carbon nanotube composites for bone tissue engineering. J Orthop Res. 2013 Sep;31(9):1374-81. doi: 10.1002/jor.22379. Epub 2013 Apr 29. PMID 23629922
- [Result] Lamplot JD, Rodeo SA, Brophy RH. A Practical Guide for the Current Use of Biologic Therapies in Sports Medicine. Am J Sports Med. 2020 Feb;48(2):488-503. doi: 10.1177/0363546519836090. Epub 2019 Apr 30. PMID 31038990
- [Result] Rodriguez HC, Gupta M, Cavazos-Escobar E, El-Amin SF 3rd, Gupta A. Umbilical cord: an allogenic tissue for potential treatment of COVID-19. Hum Cell. 2021 Jan;34(1):1-13. doi: 10.1007/s13577-020-00444-5. Epub 2020 Oct 9. PMID 33033884
- [Result] Gupta A, Cady C, Fauser AM, Rodriguez HC, Mistovich RJ, Potty AGR, Maffulli N. Cell-free Stem Cell-Derived Extract Formulation for Regenerative Medicine Applications. Int J Mol Sci. 2020 Dec 9;21(24):9364. doi: 10.3390/ijms21249364. PMID 33316880
- [Result] Main BJ, Maffulli N, Valk JA, Rodriguez HC, Gupta M, El-Amin SF 3rd, Gupta A. Umbilical Cord-Derived Wharton's Jelly for Regenerative Medicine Applications: A Systematic Review. Pharmaceuticals (Basel). 2021 Oct 27;14(11):1090. doi: 10.3390/ph14111090. PMID 34832872
- [Result] Gupta A, El-Amin SF 3rd, Levy HJ, Sze-Tu R, Ibim SE, Maffulli N. Umbilical cord-derived Wharton's jelly for regenerative medicine applications. J Orthop Surg Res. 2020 Feb 13;15(1):49. doi: 10.1186/s13018-020-1553-7. PMID 32054483
- [Result] Dernek B, Duymus TM, Koseoglu PK, Aydin T, Kesiktas FN, Aksoy C, Mutlu S. Efficacy of single-dose hyaluronic acid products with two different structures in patients with early-stage knee osteoarthritis. J Phys Ther Sci. 2016 Nov;28(11):3036-3040. doi: 10.1589/jpts.28.3036. Epub 2016 Nov 29. PMID 27942115